CLINICAL TRIAL: NCT06569823
Title: A Phase 1/2 Randomized, Observer-Blinded, Active-Controlled, Dose, Escalation Multicenter Trial to Evaluate the Safety, Tolerability, and Immunogenicity of an Investigational Herpes Zoster Vaccine (Z-1018) Compared to Shingrix® in Healthy Adult Participants 50 Years of Age and Over
Brief Title: Safety and Immunogenicity of an Investigational Herpes Zoster Vaccine (Z-1018) Compared to Shingrix® in Healthy Adults 50 Years of Age and Over
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DV2-ZOS-02
Record Dates: First submitted 2024-07-08; First posted 2024-08-26 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Shingles; Herpes Zoster; Vaccine-Preventable Diseases
MeSH Terms: conditions — Herpes Zoster; Vaccine-Preventable Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Z-1018 A1 (Part 1) (Experimental): Participants will receive a dose of Z-1018 by intramuscular (IM) injection on Day 1 and Day 85.
  Interventions: Biological: Z-1018
- Z-1018 A2 (Part 1) (Experimental): Participants will receive a dose of Z-1018 by intramuscular (IM) injection on Day 1 and Day 85.
  Interventions: Biological: Z-1018
- Z-1018 B1(a) (Part 1) (Experimental): Participants will receive a dose of Z-1018 by intramuscular (IM) injection on Day 1 and Day 57.
  Interventions: Biological: Z-1018
- Z-1018 B2(a) (Part 1 and Part 2) (Experimental): Participants will receive a dose of Z-1018 by intramuscular (IM) injection on Day 1 and Day 57.
  Interventions: Biological: Z-1018
- Z-1018 B1(b) (Part 1) (Experimental): Participants will receive a dose of Z-1018 by intramuscular (IM) injection on Day 1 and Day 85
  Interventions: Biological: Z-1018
- Z-1018 B2(b) (Part 1) (Experimental): Participants will receive a dose of Z-1018 by intramuscular (IM) injection on Day 1 and Day 85
  Interventions: Biological: Z-1018
- Z-1018 Formulation C1(a) (Part 1) (Experimental): Participants will receive a dose of Z-1018 by intramuscular (IM) injection on Day 1 and Day 57.
  Interventions: Biological: Z-1018
- Z-1018 Formulation C2(a) (Part 1) (Experimental): Participants will receive a dose of Z-1018 by intramuscular (IM) injection on Day 1 and Day 57.
  Interventions: Biological: Z-1018
- Z-1018 Formulation C1(b) (Part 1) (Experimental): Participants will receive a dose of Z-1018 by intramuscular (IM) injection on Day 1 and Day 85.
  Interventions: Biological: Z-1018
- Z-1018 Formulation C2(b) (Part 1) (Experimental): Participants will receive a dose of Z-1018 by intramuscular (IM) injection on Day 1 and Day 85.
  Interventions: Biological: Z-1018
- Shingrix (Part 1 and Part 2) (Experimental): Participants will receive a dose of Shingrix by intramuscular (IM) injection on Day 1 and Day 57, or Day 1 and Day 85.
  Interventions: Biological: Shingrix

INTERVENTIONS:
Biological: Z-1018 — Formulation for injection
  Arms: Z-1018 A1 (Part 1); Z-1018 A2 (Part 1); Z-1018 B1(a) (Part 1); Z-1018 B1(b) (Part 1); Z-1018 B2(a) (Part 1 and Part 2); Z-1018 B2(b) (Part 1); Z-1018 Formulation C1(a) (Part 1); Z-1018 Formulation C1(b) (Part 1); Z-1018 Formulation C2(a) (Part 1); Z-1018 Formulation C2(b) (Part 1)
Biological: Shingrix — Formulation for injection
  Arms: Shingrix (Part 1 and Part 2)

SUMMARY:
This is a randomized, active-controlled, observer-blinded, dose-escalation multi-center trial of 2 doses of an investigational HZ vaccine (Z-1018) in approximately 764 healthy adults.

DETAILED DESCRIPTION:
Part 1 will enroll approximately 440 participants 50 through 69 years of age (YOA) [inclusive] to 1 of 10 arms of Z-1018 or to Shingrix.

Part 2 will enroll approximately 324 participants ≥ 70 YOA to 1 arm of Z-1018 (selected from Part 1) to be administered in a 1:1 randomization ratio with Shingrix. Part 2 only: after completing the 12-month post-vaccination visit, Part 2 participants will be followed for an additional 4 years for immunopersistence and for herpes zoster (HZ) and post herpetic neuralgia (PHN).

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate; informed consent provided for the study
2. Male or female ≥ 50 years of age (Part 1: 50 through 69 years of age, inclusive; Part 2: ≥ 70 years of age
3. In good health in the opinion of the investigator, based upon medical history, physical examination, and laboratory evaluation
4. Able to comprehend and follow all required trial procedures and be available for all visits scheduled in the trial
5. Seronegative for human immunodeficiency virus (HIV), hepatitis B virus (HBV), and hepatitis C virus (HCV) as assessed during Screening
6. If female of child-bearing potential and heterosexually active, has practiced adequate contraception for at least 28 days prior to vaccination, has negative pregnancy tests just prior to vaccination, and has agreed to continue adequate contraception through 3 months following the final study injection.

Exclusion Criteria:

1. History of HZ
2. Previous vaccination against varicella (chicken pox) or HZ
3. Febrile illness within 7 days of the first trial injection (defined as at least 1 measured body temperature of ≥ 38°C, regardless of route of measurement)
4. Confirmed SARS-CoV-2/COVID-19 infection as assessed during Screening within 7 days of first trial injection.
5. If female of childbearing potential, is pregnant (known before or established at the time of screening), breastfeeding, or planning a pregnancy or to breastfeed
6. Known or suspected immunodeficiency (including but not limited to HIV/AIDS), or immunocompromised state, as assessed by medical history, past or current laboratory studies, and/or physical examination
7. History of sensitivity to any component of the trial vaccines
8. Has received the following prior to Day 1 trial injection:

   a) ≤ 14 days: i) Any licensed or authorized inactivated vaccines (including vaccines containing mRNA or CpG)

   b) ≤ 28 days: i) Any live vaccine ii) Systemic corticosteroids (≥ 20 mg/ day of prednisone or equivalent for more than 14 consecutive days) or other immunomodulators or immune suppressive medication, with the exception of inhaled steroids iii) Any investigational medicinal agent

   c) ≤ 90 days: i) Granulocyte or granulocyte-macrophage colony-stimulating factor ii) Immunoglobulins or any blood products (receipt of certain monoclonal antibodies may on a case-by-case basis be non-exclusionary if approved via consultation with Sponsor Medical Monitor) iii) Antisense oligonucleotides iv) Drugs/investigational agents with very long half-lives (defined as ≥ 60 days) (eg, radioactive iodine-125, amiodarone, nirsevimab, and evinacumab) v) Infusion of blood products

   d) ≤ 6 months before Day 1 (or likely to require during the trial period): i) chronic administration of immunosuppressants or other immune-modifying drugs

   e) At any time: DNA plasmids or other genetic therapy intended to integrate permanently into host cells
9. Is undergoing chemotherapy or expected to receive chemotherapy during the trial period; and/or has a diagnosis of cancer within the last 5 years other than squamous cell or basal cell carcinoma of the skin
10. History or current evidence of any condition, therapy, laboratory abnormality, or other finding that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
11. Underlying chronic medical condition requiring ongoing follow-up and monitoring by a healthcare provider that might affect the immune response to vaccine (eg, diabetes mellitus, chronic kidney disease)
12. Known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial
13. Current or historical autoimmune disease
14. Any skin condition and/or tattoo on both arms that may interfere with the evaluation of safety at the injection site, in the opinion of the treating investigator
15. Any other finding that the Investigator considers will make the participant unsuitable for the trial or unable to comply with the trial requirements

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 764 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Part 1 and Part 2: Percentage of participants with solicited local and systemic post-injection reactions (PIRs) | Up to 7 days following each dose
  Solicited local and systemic post-injection reactions (PIRs)
Part 1 and Part 2: Percentage of participants with Adverse events (AEs) | 28 days following each dose
  Adverse events (AEs)
Part 1 and Part 2: Percentage of participants with serious adverse events (SAEs), medically-attended adverse events (MAEs), and immune-mediated adverse events of special interest (imAESIs) | Day 1 through 12 months after the last dose of study injection
  Serious adverse events (SAEs) Medically-attended adverse events (MAEs) Immune-mediated adverse events of special interest (imAESIs)
Part 2: Vaccine response | 4 weeks after the second study injection
  Composite vaccine response rate in glycoprotein E (gE) -specific CD4+ T cells and anti-gE IgG antibodies in the Per Protocol (PP) population
Part 2: Anti-gE IgG antibody concentration | 4 weeks after the second study injection
  Geometric mean concentration (GMC) and geometric mean ratio of IgG antibodies to varicella-zoster virus (VZV) antigen-gE in the Per Protocol (PP) population

SECONDARY OUTCOMES:
Part 1: GMC of IgG antibodies to VZV antigen-gE 4 weeks after the second study injection | 4 weeks after the second study injection
  GMC to VZV gE in the Per Protocol (PP) population
Part 1: Geometric mean ratio (GMR) of IgG antibodies to VZV antigen gE | 4 weeks after the second study injection
  Geometric mean ratio (GMR) of IgG antibodies to VZV antigen gE in the Per Protocol (PP) population
Part 1: Geometric mean fold increase (GMFI) of IgG antibodies to VZV antigen gE | 4 weeks after the second study injection
  Geometric mean fold increase (GMFI) of IgG antibodies to VZV antigen gE in the Per Protocol (PP) population
Part 1 and Part 2: Vaccine response rate (VRR) for anti-gE IgG antibodies to VZV antigen gE | 4 weeks after the second study injection
  Vaccine response rate (VRR) for anti-gE IgG antibodies to VZV antigen gE in the Per Protocol (PP) population
Part 2: VRR for gE-specific CD4+ T cells | 4 weeks after second study injection
  VRR for gE-specific CD4+ T cells in the Per Protocol (PP) population

CONTACTS AND LOCATIONS:
Overall Officials: Robert Janssen, MD, Study Chair — Dynavax Technologies Corporation
Locations (13):
- Australia (10):
  - Emeritus Research, Botany, New South Wales
  - Canopy Clinical Northern Beaches, Brookvale, New South Wales
  - Paratus Clinical Research Central Coast, Kanwal, New South Wales
  - Sutherland Shire Clinical Research, Miranda, New South Wales
  - Innovate Clinical Research, Waitara, New South Wales
  - Canopy Clinical Wollongong, Wollongong, New South Wales
  - Paratus Clinical Research Brisbane, Herston, Queensland
  - Momentum Clinical Research Wellers Hill, Tarragindi, Queensland
  - Veritus Research, Bayswater, Victoria
  - Emeritus Research, Camberwell, Victoria
- New Zealand (3):
  - Optimal Clinical Trials Ltd - North, Auckland
  - Optimal Clinical Trials Ltd - Central, Auckland
  - Momentum Wellington, Wellington

IPD SHARING:
Plan to Share IPD: No